CLINICAL TRIAL: NCT07150663
Title: A Prospective, Randomized, Parallel-Controlled Clinical Study of Nanocrystalline Megestrol Acetate in Concurrent Chemoradiotherapy for Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Nanocrystalline Megestrol Acetate in Concurrent Chemoradiotherapy for Locally Advanced Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Megaxia CRT-NSCLC-01
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nanocrystalline Megestrol Acetate Oral Suspension+ Standard Therapy (Experimental)
  Interventions: Drug: Nano-crystalline Megestrol Acetate Oral Suspension; Other: Standard Therapy
- Placebo+ Standard Therapy (Placebo Comparator)
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Drug: Nano-crystalline Megestrol Acetate Oral Suspension — Nanocrystalline Megestrol Acetate Oral Suspension Nanocrystalline Megestrol Acetate Oral Suspension (125 mg/mL) was administered to the study group at 5 mL orally once daily (equivalent to 625 mg/day) until disease progression or completion of 8 weeks (maximum treatment duration: 8 weeks), whichever occurred first.
  Arms: Nanocrystalline Megestrol Acetate Oral Suspension+ Standard Therapy
Other: Standard Therapy — Standard Therapy

SUMMARY:
This study is a prospective, randomized, parallel-controlled clinical trial, primarily aimed at evaluating the efficacy and safety of Nanocrystalline Megestrol Acetate combined with standard therapy, compared with placebo combined with standard therapy, in improving appetite and body weight during concurrent chemoradiotherapy for patients with locally advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent (ICF).
2. Age ≥ 18 years at enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
4. Expected survival ≥ 6 months.
5. Histologically or cytologically confirmed, unresectable or inoperable locally advanced (stage III) non-small cell lung cancer (adenocarcinoma or squamous cell carcinoma) according to the 8th edition of the TNM classification by the International Association for the Study of Lung Cancer (IASLC) and the American Joint Committee on Cancer (AJCC).
6. Planned to receive radical concurrent chemoradiotherapy.
7. Body mass index (BMI) ≤ 25.
8. At least one measurable tumor lesion according to RECIST v1.1.

Exclusion Criteria:

1. Presence of any condition affecting gastrointestinal absorption, such as difficulty swallowing, malabsorption, or uncontrollable vomiting; currently receiving tube feeding or parenteral nutrition; suffering from anorexia due to neurological or psychiatric disorders, or difficulty eating due to pain.
2. Currently taking or planning to take other medications that increase appetite or body weight, such as corticosteroids (excluding short-term dexamethasone during chemotherapy), androgens, progestins, thalidomide, olanzapine, anamorelin, or other appetite stimulants.
3. Patients with Cushing's syndrome, adrenal or pituitary insufficiency; patients with poorly controlled diabetes.
4. Postmenopausal women with a history of abnormal vaginal bleeding within one year; premenopausal women with a history of abnormal endometrial thickening (>15 mm) within one year.
5. Current radiological or clinical evidence of gastrointestinal obstruction.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of appetite decrease assessed by A/CS-12 (Anorexia/Cachexia Subscale of Functional Assessment of Anorexia/Cachexia Therapy) | over an 8-week period
Proportion of individuals with weight loss exceeding 5% relative to baseline | over an 8-week period

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, TongjiMedical College, Huazhong University of Science and Technology, Wuhan, Hubei, China